CLINICAL TRIAL: NCT03614520
Title: Evaluation of Bioavailability and Metabolism of Diet Phenolic Compounds
Acronym: dopet4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Rafael de la Torre, Director of the Neurosciences Department in IMIM, Parc de Salut Mar
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IMIMFTCL/DOPET4
Record Dates: First submitted 2018-07-10; First posted 2018-08-03 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — Olive Oil; Water; Ethanol

STUDY DESIGN:
Intervention Model Description: A 40 people group of healthy men and women. Two Cohorts group of 20 healthy volunteers of both genders.
Masking Description: The subjects, because of the wine taste that cannot be hidden, will know what they drink, except from the three beers (the three types will not be distinguishable).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub-study A : olive oil, wine, both, or water (placebo). (Experimental): After being selected, subjects will do 4 experimental sessions (each separated by 3 days minimum) in which ones they will drink olive oil, red wine, red wine and olive oil, or water (placebo). The order of the experimental sessions will be drawn.
  Interventions: Other: Administration of olive oil; Other: Administration of red wine; Other: Combination of red wine and olive oil; Other: Water
- Sub-study B : three types of beer, and wine (Experimental): The subjects will do 4 experimental sessions (each separated by 3 days minimum) in wich ones they will drink a beer (250mL) or wine (150mL). The order of the experimental sessions will be drawn.
  Interventions: Other: Administration of red wine; Other: Dark beer; Other: Light Beer; Other: Alcohol free Beer

INTERVENTIONS:
Other: Administration of olive oil — 25 mL of extra virgin olive oil
  Arms: Sub-study A : olive oil, wine, both, or water (placebo).
Other: Administration of red wine — 150 mL or Red Wine
Other: Combination of red wine and olive oil — 150 mL of Red wine + 25 mL of Extra Virgin Olive oil will be administred at the same time
  Arms: Sub-study A : olive oil, wine, both, or water (placebo).
Other: Water — Mineral water will be given as placebo
  Arms: Sub-study A : olive oil, wine, both, or water (placebo).
Other: Dark beer — 250 mL of IPA beer (alcohol 8.5% vol)
  Arms: Sub-study B : three types of beer, and wine
Other: Light Beer — 250 mL of blonde ale beer (alcohol 4,5% vol)
  Arms: Sub-study B : three types of beer, and wine
Other: Alcohol free Beer — 250 mL of alcohol free beer (alcohol 0.0% vol)
  Arms: Sub-study B : three types of beer, and wine

SUMMARY:
This study aims at studying in depth the absorption and metabolism of phenolic compounds of olive oil, wine and beer. This study is divided into 2 sub-studies in order to evaluate each one of the objectives.

DETAILED DESCRIPTION:
The study is divided in two sub-studies to explore each objective.

One the one hand, a group of people will drink olive oil, or wine, or both. This is done to see if combining these two drinks will improve the absorption and bioavailibility of phenolic compounds that they contain, promoting by synergy their antioxidant activity at a postprandial level. The main compounds studied are the Resveratrol (RSVT), the Hydroxytyrosol (HT), tyrosol (TIR) and their metabolits.

One the other hand, an group of people will drink 3 different beers ( with 3 different degrees of alcohol), or wine, in order to study the absorption of TIR in relation to the alcohol degree. It also aims at assessing if the gas contained in beer contributes to TIR absorption.

At different times after the administration of drinks, urine and blood samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Men and women from 18 to 45 years old.
* Understand and accepting the procedures of the trial and sign an informed consent.
* Have a history and physical exams that show that there is no organic issue, and an analysis and ECG in the normal limits.
* Have an BMI between 18.5 and 30 kg/m2.
* caucasian race

Exclusion Criteria:

* Smokers
* Persons with chronical disease
* Persons with BMI>30 or <18.5 kg/m2.
* Persons with history of multiple allergies or obvious intestinal, hepatic, renal issues or other problems that could suppose a deterioration of absorption, distribution or metabolism of polyphenols.
* Persons who take anti-oxidant products, including vitamins, herbal medication or dietetics complementation that could interfere in the study objectives.
* Persons with restrictive diet (including vegetarian diet).
* Persons with history of hypersensibility or intolerance to alcohol.
* Persons with a daily consumption of alcohol >50g or who have consumed illegal drug in the month preceding the study.
* Persons who have participated in an other clinical trial the month preceding the study.
* Persons who have done a blood donation during the last 3 months before the beginning of the study (only appliable to the subjects of A sub-study).
* Persons who have a positive serology for B or C hepatitis or HIV.
* Pregnant or breastfeeding women, or any other situation prohibiting alcohol consumption.
* Persons who have consummed NSAIDs (especially acetylsalicylic acid) or antioxidants or vitamin complementation, during the 2 weeks preceding the beginning of the study.
* Illiterate persons

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Sub-study A : Basal dosing of urinary phenolic compounds and their metabolites concentrations | 2 hours before administration to administration (-2 to 0 hours)
Sub-study A : Basal dosing of urinary phenolic compounds and their metabolites concentrations | 0-2 hours; 2-4 hours; 4-6 hours; 6-12 hours; 12-24 hours post administration
Sub-study A : Postprandial dosing of plasmatic phenolic compounds and their metabolites concentrations | baseline, 30 minutes; 45 minutes; 1 hours; 1.5 hours; 2 hours; 6 hours post administration
Sub-study B : Basal dosing of urinary phenolic compounds and their metabolites concentrations | 2 hours before administration to administration (-2 to 0 hours)
Sub-study B : Postprandial dosing of urinary phenolic compounds and their metabolites concentrations | 0-2 hours; 2-4 hours; 4-6 hours; 6-12 hours; 12-24 hours

SECONDARY OUTCOMES:
Sub-study A : Postprandial dosing of plasmatic glucose | baseline, 30 minutes; 45 minutes; 1 hours; 1.5 hours; 2 hours; 6 hours post administration
Sub-study A : Postprandial dosing of plasmatic insulin | baseline, 30 minutes; 45 minutes; 1 hours; 1.5 hours; 2 hours; 6 hours post administration
Sub-study A : Postprandial dosing of plasmatic total cholesterol | baseline, 30 minutes; 45 minutes; 1 hours; 1.5 hours; 2 hours; 6 hours post administration
Sub-study A : Postprandial dosing of plasmatic triglyceride | baseline, 30 minutes; 45 minutes; 1 hours; 1.5 hours; 2 hours; 6 hours post administration
Sub-study A : Postprandial dosing of plasmatic LDL | baseline, 30 minutes; 45 minutes; 1 hours; 1.5 hours; 2 hours; 6 hours post administration
Sub-study A : Postprandial dosing of plasmatic oxidated-LDL | baseline, 30 minutes; 45 minutes; 1 hours; 1.5 hours; 2 hours; 6 hours post administration
Sub-study A : Postprandial dosing of plasmatic HDL concentrations. | baseline, 30 minutes; 45 minutes; 1 hours; 1.5 hours; 2 hours; 6 hours post administration
Sub-study A : Basal cardiovascular activity : blood pressure | 15 minutes before administration
Sub-study A : Basal cardiovascular activity: heart rate | 15 minutes before administration
Sub-study A : Basal cardiovascular activity : endothelial function. | 15 minutes before administration
  Endothelial function will be assessed as flow-mediated dilation using endoPAT 2000 (Itamar Medical device). Flow-mediated dilation is the most widely used method to test endothelial function since it is non-invasive, and measures by ultrasounds the response to increased shear stress, commonly in the brachial artery
Sub-study A : Postprandial cardiovascular activity : blood pressure | 1 hour and 2 hours post administration
Sub-study A : Postprandial cardiovascular activity : heart rate | 1 hour and 2 hours post administration
Sub-study A : Postprandial cardiovascular activity: endothelial function. | 1 hour and 2 hours post administration
  Endothelial function will be assessed as flow-mediated dilation using endoPAT 2000 (Itamar Medical device). Flow-mediated dilation is the most widely used method to test endothelial function since it is non-invasive, and measures by ultrasounds the response to increased shear stress, commonly in the brachial artery
Sub-study B : Basal cardiovascular activity : blood pressure | 15 minutes before administration
Sub-study B : Basal cardiovascular activity: heart rate. | 15 minutes before administration
Sub-study B : Postprandial cardiovascular activity : blood pressure | 30 minutes, 1hour, 2 hours and 4 hours post administration
Sub-study B : Postprandial cardiovascular activity: heart rate. | 30 minutes, 1hour, 2 hours and 4 hours post administration
Sub-study B : Concentration of alcohol in the exhaled breath | 15 minutes before administration
  Blood alcohol (ethanol) concentration is correlated with the concentration of alcohol in the exhaled breath at end-exhalation (BrAC). It is a non-invasive method that has been used to quantify alcohol intake.
Sub-study B : Postprandial Concentration of alcohol in the exhaled breath | 30 minutes, 1hour, 2 hours and 4 hours post administration
  Blood alcohol (ethanol) concentration is correlated with the concentration of alcohol in the exhaled breath at end-exhalation (BrAC). It is a non-invasive method that has been used to quantify alcohol intake.
Sub-study B : Basal isoxanthohumol urinary concentration | 2 hours before administration to administration (-2 to 0 hours)
  Isoxanthohumol is a biomarker of beer consumption.
Sub-study B : Postprandial isoxanthohumol urinary concentration | 0-2 hours; 2-4 hours; 4-6 hours; 6-12 hours; 12-24 hours post administration
  Isoxanthohumol is a biomarker of beer consumption.
Sub-study B : Basal urinary creatinine concentration | 2 hours before administration to administration (-2 to 0 hours)
Sub-study B : Basal urinary urinary pH. | 2 hours before administration to administration (-2 to 0 hours)
  pH is a logarithmic scale used to specify the acidity or basicity of an aqueous solution.
Sub-study B : Postprandial urinary creatinine concentration | 0-2 hours; 2-4 hours; 4-6 hours; 6-12 hours; 12-24 hours post administration
Sub-study B : Postprandial urinary urinary pH. | 0-2 hours; 2-4 hours; 4-6 hours; 6-12 hours; 12-24 hours post administration
  pH is a logarithmic scale used to specify the acidity or basicity of an aqueous solution.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael de la Torre Fornell, Dr, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- Consorci Parc de Salut Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu L, Sun D. Adherence to Mediterranean diet and risk of developing cognitive disorders: An updated systematic review and meta-analysis of prospective cohort studies. Sci Rep. 2017 Jan 23;7:41317. doi: 10.1038/srep41317. PMID 28112268
- [Background] Rodriguez-Morato J, Robledo P, Tanner JA, Boronat A, Perez-Mana C, Oliver Chen CY, Tyndale RF, de la Torre R. CYP2D6 and CYP2A6 biotransform dietary tyrosol into hydroxytyrosol. Food Chem. 2017 Feb 15;217:716-725. doi: 10.1016/j.foodchem.2016.09.026. Epub 2016 Sep 7. PMID 27664690
- [Background] Perez-Mana C, Farre M, Rodriguez-Morato J, Papaseit E, Pujadas M, Fito M, Robledo P, Covas MI, Cheynier V, Meudec E, Escudier JL, de la Torre R. Moderate consumption of wine, through both its phenolic compounds and alcohol content, promotes hydroxytyrosol endogenous generation in humans. A randomized controlled trial. Mol Nutr Food Res. 2015 Jun;59(6):1213-6. doi: 10.1002/mnfr.201400842. Epub 2015 Apr 27. PMID 25712532
- [Background] Granados-Principal S, Quiles JL, Ramirez-Tortosa CL, Sanchez-Rovira P, Ramirez-Tortosa MC. Hydroxytyrosol: from laboratory investigations to future clinical trials. Nutr Rev. 2010 Apr;68(4):191-206. doi: 10.1111/j.1753-4887.2010.00278.x. PMID 20416016
- [Background] Oliveras-Lopez MJ, Molina JJ, Mir MV, Rey EF, Martin F, de la Serrana HL. Extra virgin olive oil (EVOO) consumption and antioxidant status in healthy institutionalized elderly humans. Arch Gerontol Geriatr. 2013 Sep-Oct;57(2):234-42. doi: 10.1016/j.archger.2013.04.002. Epub 2013 May 1. PMID 23642776
- [Background] Weinbrenner T, Fito M, de la Torre R, Saez GT, Rijken P, Tormos C, Coolen S, Albaladejo MF, Abanades S, Schroder H, Marrugat J, Covas MI. Olive oils high in phenolic compounds modulate oxidative/antioxidative status in men. J Nutr. 2004 Sep;134(9):2314-21. doi: 10.1093/jn/134.9.2314. PMID 15333722
- [Background] Castaner O, Covas MI, Khymenets O, Nyyssonen K, Konstantinidou V, Zunft HF, de la Torre R, Munoz-Aguayo D, Vila J, Fito M. Protection of LDL from oxidation by olive oil polyphenols is associated with a downregulation of CD40-ligand expression and its downstream products in vivo in humans. Am J Clin Nutr. 2012 May;95(5):1238-44. doi: 10.3945/ajcn.111.029207. Epub 2012 Mar 21. PMID 22440854
- [Background] Hernaez A, Fernandez-Castillejo S, Farras M, Catalan U, Subirana I, Montes R, Sola R, Munoz-Aguayo D, Gelabert-Gorgues A, Diaz-Gil O, Nyyssonen K, Zunft HJ, de la Torre R, Martin-Pelaez S, Pedret A, Remaley AT, Covas MI, Fito M. Olive oil polyphenols enhance high-density lipoprotein function in humans: a randomized controlled trial. Arterioscler Thromb Vasc Biol. 2014 Sep;34(9):2115-9. doi: 10.1161/ATVBAHA.114.303374. Epub 2014 Jul 24. PMID 25060792
- [Background] Ruano J, Lopez-Miranda J, de la Torre R, Delgado-Lista J, Fernandez J, Caballero J, Covas MI, Jimenez Y, Perez-Martinez P, Marin C, Fuentes F, Perez-Jimenez F. Intake of phenol-rich virgin olive oil improves the postprandial prothrombotic profile in hypercholesterolemic patients. Am J Clin Nutr. 2007 Aug;86(2):341-6. doi: 10.1093/ajcn/86.2.341. PMID 17684203
- [Background] Ruano J, Lopez-Miranda J, Fuentes F, Moreno JA, Bellido C, Perez-Martinez P, Lozano A, Gomez P, Jimenez Y, Perez Jimenez F. Phenolic content of virgin olive oil improves ischemic reactive hyperemia in hypercholesterolemic patients. J Am Coll Cardiol. 2005 Nov 15;46(10):1864-8. doi: 10.1016/j.jacc.2005.06.078. Epub 2005 Oct 24. PMID 16286173
- [Background] De la Torre R, Corella D, Castaner O, Martinez-Gonzalez MA, Salas-Salvado J, Vila J, Estruch R, Sorli JV, Aros F, Fiol M, Ros E, Serra-Majem L, Pinto X, Gomez-Gracia E, Lapetra J, Ruiz-Canela M, Basora J, Asensio EM, Covas MI, Fito M. Protective effect of homovanillyl alcohol on cardiovascular disease and total mortality: virgin olive oil, wine, and catechol-methylation. Am J Clin Nutr. 2017 Jun;105(6):1297-1304. doi: 10.3945/ajcn.116.145813. Epub 2017 Apr 26. PMID 28446500